CLINICAL TRIAL: NCT06583161
Title: Emulation of the Moderate Alcohol and Cardiovascular Health Trial (MACH15)
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Goodarz Danaei, Professor, Harvard School of Public Health (HSPH)
Other Study IDs: IRB23-1533
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Infarction; Ischemic Stroke; Angina Pectoris; Coronary Revascularization; All-cause Mortality; Cardiovascular Death; Type 2 Diabetes; Heart Failure; Atrial Fibrillation; Cancer; Dementia; Depression; Infections; Injuries; Liver Cirrhosis
MeSH Terms: conditions — Myocardial Infarction; Ischemic Stroke; Angina Pectoris; Diabetes Mellitus, Type 2; Heart Failure; Atrial Fibrillation; Neoplasms; Dementia; Depression; Infections; Wounds and Injuries; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Moderate drinkers: Participants who report drinking up to 16 grams of alcohol daily or almost daily on a repeated assessment center visit, or who report drinking 8-16 grams of alcohol 4 or more times per week on the web-based mental health questionnaire.
  Interventions: Behavioral: Moderate drinking
- Quitters: Participants who report not drinking alcohol on a repeated assessment center visit or in the web-based mental health questionnaire.
  Interventions: Behavioral: Quitting
- Social drinkers: Participants who report drinking up to 16 grams of alcohol 1-2 days per week or drinking 1-3 times per month or only on special occasions on a repeated assessment center visit, or who report drinking 8-16 grams of alcohol 2-3 times per week or drinking 4 times per month or less in the web-based mental health questionnaire.
  Interventions: Behavioral: Social drinking
- Heavy/binge drinkers: Participants who report drinking more than 16 grams of alcohol daily or almost daily or drinking more than 40 grams of alcohol 1-2 days per week on a repeated assessment center visit, or who report drinking 24 grams of alcohol or more 4 or more times per week or 40 grams of alcohol or more 2-3 times per week on the web-based mental health questionnaire.
  Interventions: Behavioral: Heavy/binge drinking

INTERVENTIONS:
Behavioral: Moderate drinking — Drink up to 16 grams of alcohol daily or almost daily [repeated assessment center visit] or 8-16 grams of alcohol 4 or more times per week [web-based mental health questionnaire]
  Groups: Moderate drinkers
Behavioral: Quitting — No alcohol consumption
  Groups: Quitters
Behavioral: Social drinking — Drink up to 16 grams of alcohol 1-2 days per week or drink 1-3 times per month or only on special occasions [repeated assessment center visit], or drink 8-16 grams of alcohol 2-3 times per week or drink 4 times per month or less [web-based mental health questionnaire]
  Groups: Social drinkers
Behavioral: Heavy/binge drinking — Drink more than 16 grams of alcohol daily or almost daily or more than 40 grams of alcohol 1-2 days per week [repeated assessment center visit], or 24 grams of alcohol or more 4 or more times per week or 40 grams of alcohol or more 2-3 times per week [web-based mental health questionnaire]
  Groups: Heavy/binge drinkers

SUMMARY:
The aim of this study is to assess how long-term alcohol consumption influences health risks by emulating the Moderate Alcohol and Cardiovascular Health Trial (MACH15). In the first step, the protocol of the emulation of MACH15, including eligibility criteria, alcohol regimens and assignment, follow-up, endpoints, causal contrasts of interest, and statistical analysis was specified. In the second step, the investigators will emulate an adapted version of MACH15 following the specified protocol using data from the UK Biobank.

DETAILED DESCRIPTION:
Observational data suggests that alcohol consumption lowers the risk of cardiovascular disease (CVD) compared to no consumption. Whether this relationship is truly causal remains uncertain because of the inherent limitations of observational studies, including unmeasured confounding and reverse causation. Mendelian randomization studies using genes as instrumental variables for alcohol are partially protected from these biases and have found no or harmful associations between alcohol consumption and CVD.

To date, there has only been one long-term randomized controlled trial to investigate the cardiovascular effects of alcohol consumption: the Moderate Alcohol and Cardiovascular Health Trial (MACH15; NCT Number: NCT03169530). It was, however, terminated shortly after initiation. An alternative to a real randomized trial like MACH15, which must first be completed and is subject to strict eligibility criteria to ensure safety, is to use observational data to emulate a (hypothetical) pragmatic randomized trial.

In this study, the investigators will emulate an adapted version of MACH15 using observational data from the UK Biobank, a large prospective cohort study of over 500,000 participants. The cardiometabolic effects of moderate drinking vs quitting, as originally planned in MACH15, as well as the effects of social and heavy/binge drinking on CVD, type 2 diabetes, other alcohol-related health outcomes, and death will be quantified.

ELIGIBILITY:
Inclusion criteria:

* 40-69 years old at enrollment
* Currently drinking

Exclusion criteria:

* Within the six months prior to baseline, cardiovascular disease event (myocardial infarction, revascularization procedure, or stroke)
* Hospitalization due to heart failure
* History of any of the following alcohol-related conditions, confirmed by a hospital record: alcoholic cardiomyopathy, alcoholic gastritis, alcoholic liver disease, degeneration of the nervous system due to alcohol, alcoholic myopathy, alcoholic polyneuropathy, alcohol-induced acute or chronic pancreatitis, alcohol use disorder; or self-reported history of alcoholic liver disease or alcohol use disorder
* Dual antiplatelet therapy or coumarin anticoagulants
* Serious chronic liver disease (active hepatitis B or C infection) in the past 6 months before baseline
* Personal history of any colon or liver cancer
* Personal history of breast cancer
* Diagnosis of dementia
* Not willing or able to provide a signed and dated informed consent form
* Reduced alcohol compared to 10 years ago due to illness, ill health, or doctor's advice
* Self-reported poor health

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All people aged 40-69 years who were registered with the National Health Service and lived within 25 miles of one of the 22 study assessment centers in England, Wales, and Scotland were invited to participate. Overall, about 9.2 million invitations were mailed in order to recruit 503,325 participants (i.e. a response rate of 5.47%)
Sampling Method: Non-Probability Sample
Enrollment: 503325 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease or death | From date of baseline measurement until the date of first cardiovascular disease or death documented in hospital or death registry data, administrative censoring, or loss to follow-up, whichever came first, assessed up to 200 months
  Composite endpoint comprised of the first occurrence of a non-fatal myocardial infarction, non-fatal ischemic stroke, hospitalization for angina, coronary/carotid revascularization, and all-cause mortality

SECONDARY OUTCOMES:
Cardiovascular disease | From date of baseline measurement until the date of first cardiovascular disease documented in hospital or death registry data, administrative censoring, loss to follow-up, or death from other causes, whichever came first, assessed up to 200 months
  Composite endpoint comprised of the first occurrence of a non-fatal myocardial infarction, non-fatal ischemic stroke, hospitalization for angina, coronary/carotid revascularization, and cardiovascular death
Type 2 diabetes | From date of baseline measurement until the date of first type 2 diabetes documented in hospital or death registry data, administrative censoring, loss to follow-up, or death from other causes, whichever came first, assessed up to 200 months
  Progression among normoglycemic and pre-diabetes individuals to type 2 diabetes
Alcohol-related disease or death | From date of baseline measurement until the date of first alcohol-related disease or death documented in hospital, cancer, or death registry data, administrative censoring, or loss to follow-up, whichever came first, assessed up to 200 months
  Composite endpoint comprised of the first occurrence of a non-fatal myocardial infarction, non-fatal ischemic stroke, heart failure, atrial fibrillation, cancer (except non-melanoma skin cancer), dementia, depression, infection with hospitalization, injury with hospitalization, liver cirrhosis, type 2 diabetes, and all-cause mortality

OTHER OUTCOMES:
Hard cardiovascular disease or death | From date of baseline measurement until the date of first hard cardiovascular disease or death documented in hospital or death registry data, admin. censoring, loss to follow-up, or death from other causes, whichever came first, assessed up to 200 months
  Composite endpoint comprised of the first occurrence of a non-fatal myocardial infarction, non-fatal ischemic stroke, and cardiovascular death
Cardiovascular death | From date of baseline measurement until the date of cardiovascular death documented in death registry data, administrative censoring, loss to follow-up, or death from other causes, whichever came first, assessed up to 200 months
  Cardiovascular death
Non-fatal myocardial infarction | From date of baseline measurement until the date of first non-fatal myocardial infarction documented in hospital data, administrative censoring, loss to follow-up, or death, whichever came first, assessed up to 200 months
  First occurrence of a non-fatal myocardial infarction
Non-fatal ischemic stroke | From date of baseline measurement until the date of first non-fatal ischemic stroke documented in hospital data, administrative censoring, loss to follow-up, or death, whichever came first, assessed up to 200 months
  First occurrence of a non-fatal ischemic stroke
Hospitalization for angina | From date of baseline measurement until the date of first hospitalization for angina documented in hospital data, administrative censoring, loss to follow-up, or death, whichever came first, assessed up to 200 months
  First hospitalization for angina
Coronary/carotid revascularization | From date of baseline measurement until the date of first coronary/carotid revascularization documented in hospital data, administrative censoring, loss to follow-up, or death, whichever came first, assessed up to 200 months
  First coronary/carotid revascularization
All-cause mortality | From date of baseline measurement until the date of death documented in death registry data, administrative censoring, or loss to follow-up, whichever came first, assessed up to 200 months
  Death

IPD SHARING:
Plan to Share IPD: No
Access to the UK Biobank data can be requested via the official website https://www.ukbiobank.ac.uk.

REFERENCES:
- [Background] Spiegelman D, Lovato LC, Khudyakov P, Wilkens TL, Adebamowo CA, Adebamowo SN, Appel LJ, Beulens JW, Coughlin JW, Dragsted LO, Edenberg HJ, Eriksen JN, Estruch R, Grobbee DE, Gulayin PE, Irazola V, Krystal JH, Lazo M, Murray MM, Rimm EB, Schrieks IC, Williamson JD, Mukamal KJ. The Moderate Alcohol and Cardiovascular Health Trial (MACH15): Design and methods for a randomized trial of moderate alcohol consumption and cardiometabolic risk. Eur J Prev Cardiol. 2020 Dec;27(18):1967-1982. doi: 10.1177/2047487320912376. Epub 2020 Apr 6. PMID 32250171